CLINICAL TRIAL: NCT04715282
Title: Effectiveness of the Epley Maneuver Versus Vestibular Exercises in the Treatment of Benign Paroxysmal Positional Vertigo (BPPV)
Brief Title: The Epley Maneuver Versus Cawthorne-Cooksey Exercises in the Treatment of Benign Paroxysmal Positional Vertigo (BPPV)
Acronym: BPPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Habibe Serap Inal, Prof, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstinyeU
Record Dates: First submitted 2021-01-12; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Benign Paroxysmal Positional Vertigo
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epley maneuver (Other): The Epley maneuver was performed for all patients (both EpleyM and EpleyM&Exe groups) included in this study until nystagmus had disappeared in each position. If nystagmus/vertigo was not seen, the Epley maneuver was not performed for patients at the 1st, 3rd, and 6th week assessments.
  Interventions: Procedure: Epley maneuver
- Cawthorne-Cooksey exercises combined with the Epley maneuver (Other): Additional Cawthorne-Cooksey exercises were prescribed to the EpleyM&Exe group. The physiotherapist explained and demonstrated the exercises to each patient and the patients practiced the exercises until they performed them correctly. Then the exercises were prescribed twice a day and repeated 10 times for 6 weeks as a home exercise program.
  Interventions: Procedure: Epley maneuver

INTERVENTIONS:
Procedure: Epley maneuver — Epley maneuver

SUMMARY:
Observation of the effects of Cawthorne-Cooksey exercises applied after the Epley maneuver on balance, vertigo symptoms, and quality of life in BPPV patients.

DETAILED DESCRIPTION:
Study Objective:

To observe the efficacy of Cawthorne-Cooksey exercises applied after the Epley maneuver on balance, vertigo symptoms, and quality of life in patients with posterior canal BPPV.

Study Design:

Single-blind randomized controlled study

Sample Size:

Thirty-six patients were recruited in the study and were randomized equally into Epley maneuver (EpleyM) and Epley maneuver and exercise (EpleyM&Exe) groups.

Study Method:

All patients were treated with the Epley maneuver, while CawthorneCooksey exercises were given to the EpleyM&Exe group as home exercises for 6 weeks. Static and dynamic balance, vertigo and associated symptoms, and quality of life were assessed with the Nintendo Wii Balance Board, Berg Balance Test, Vertigo Symptom Scale, and Dizziness Handicap Inventory, respectively. The assessments were repeated at the 1st, 3rd, and 6th weeks.

ELIGIBILITY:
Inclusion Criteria:

1. having posterior semicircular canal BPPV with upbeating-torsional nystagmus and positional vertigo as evaluated by the Dix-Hallpike Test
2. agreeing to undergo the Epley maneuver after that test
3. agreeing to participate in the study

Exclusion Criteria:

1. having history or symptoms of vestibular system disorders other than BPPV or central nervous system disorders causing dizziness
2. having cervical and/or lumbar pathology due to which the Epley maneuver could not be performed
3. having lower extremity pain or an operation that prevented standing and/or weight bearing
4. having anterior or horizontal canal BPPV
5. having previously undergone a vestibular rehabilitation program

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Nintendo Wii Balance Board (WBB) | one hour
  COP displacement on double leg with eyes open/closed (%): Lower scores (approaching 50%) indicate better static balance.
  Frontal plane stability on dominant leg with eyes open/closed (%): The total score ranges between 0 and 100%. Higher scores indicate better static balance.
Berg Balance Test (BBT) | one hour
  The minimum score of the BBT is 0 and the total maximum score of the BBT is 56. Higher scores indicate better dynamic balance.

SECONDARY OUTCOMES:
Vertigo Symptom Scale (VSS) | one hour
  The total score ranges between 0 and 60 points, with higher scores indicating lower vertigo associated symptoms.
Dizziness Handicap Inventory (DHI) | one hour
  The total score ranges between 0 and 100 points, with higher scores indicating lower quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ekin Taçalan, Principal Investigator — Dr. Sami Ulus Maternity, Children Health and Diseases Education and Research Hospital; H.Serap İnal, Principal Investigator — Istinye University, Faculty of Health Sciences, Physiotherapy and Rehabilitation Department

IPD SHARING:
Plan to Share IPD: No